CLINICAL TRIAL: NCT03710902
Title: Empowerment and Mobile Technology in the Control of Cardiovascular Risk Factors in Patients With Ischemic Stroke
Acronym: CARDIOSTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jukka Putaala (Other)
Responsible Party: Sponsor-Investigator, Jukka Putaala, Head of Stroke Unit, Hospital District of Helsinki and Uusimaa
Organization: Hospital District of Helsinki and Uusimaa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUS/53/2017; TYH2016127 (Other Grant/Funding Number: Hospital District of Helsinki and Uusimaa)
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack; Atrial Fibrillation; Hypertension; Empowerment
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Atrial Fibrillation; Hypertension; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical endpoints will be assessed according to PROBE principles, i.e. outcomes assessors are masked to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Diagnostic Test: ECG monitoring for 3 weeks; Other: Self-monitoring of BP and self-titration of antihypertensive medication
- Control (No Intervention): Standard diagnostic work-up, follow-up, and treatment of hypertension.

INTERVENTIONS:
Diagnostic Test: ECG monitoring for 3 weeks — A 3-week continuous ECG monitoring to detect occult AF.
  Arms: Intervention
Other: Self-monitoring of BP and self-titration of antihypertensive medication — One-week monthly self-monitoring of BP and self-titration of antihypertensive medication according to a pre-specified protocol, assisted with a mobile device application.
  Arms: Intervention

SUMMARY:
The CARDIOSTROKE is a randomized trial comparing mobile-device assisted control of hypertension together with screening of occult atrial fibrillation to standard care in patients with recent ischemic stroke or transient ischemic attack.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and hypertension are among the main treatable risk factors for ischemic stroke and transient ischemic attack (TIA). Detecting paroxysmal atrial fibrillation in stroke patients is challenging, but highly relevant since anticoagulation can effectively reduce the risk of recurrent strokes. Furthermore, hypertension remains poorly controlled even after stroke despite multiple available treatment options. In the CARDIOSTROKE trial, the investigators aim to randomize 405 patients with recent ischemic stroke or TIA into (1) standard diagnostic work-up, follow-up and treatment (control group) and (2) 3-week ECG monitoring to detect occult AF and self-monitoring of blood pressure with mobile-device-assisted self-titration of antihypertensive medication (intervention group). Randomization will occur 2:1 into control and intervention groups. The co-primary outcomes include (1) incidence of new-onset AF and (2) difference in the mean blood pressure at 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or transient ischemic attack (ABCD2 score ≥3)
* Age ≥40 years
* Pre-existing or newly diagnosed hypertension
* Informed consent from the patient or legal representative

Exclusion Criteria:

* Known high-risk source of cardioembolism
* Known indication for anticoagulation
* Contraindication for anticoagulation
* Pacemaker
* Non-compliance to study interventions as judged by the investigator
* Serious condition hampering the study conduct

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2018-10-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with New Atrial fibrillation | 12 months
  New diagnosis of atrial fibrillation (>30 s)
Change in Blood Pressure | 12 months
  Mean change in systolic/diastolic blood pressure

SECONDARY OUTCOMES:
Number of Participants with New Cardiovascular Events within 12 Months | 12 months
  Any of stroke, myocardial infarction, revascularization, or cardiovascular death
Number of Participants with New Cardiovascular Events within 36 Months | 36 months
  Any of stroke, myocardial infarction, revascularization, or cardiovascular death
Health Care Costs | 36 months
  Total direct healthcare costs

OTHER OUTCOMES:
Rate of Adverse Events | 12 months
  Adverse events related to ECG monitoring, blood pressure home monitoring, and mobile-device assisted self-adjustment of blood pressure medication according to a pre-specified protocol.
Rate of Severe Adverse Events | 12 months
  Severe adverse event related to mobile-device assisted self-adjustment of blood pressure medication according to a pre-specified protocol.

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Kanta-Häme Central Hospital, Hämeenlinna
  - Helsinki University Hospital, Helsinki
  - Hyvinkää Hospital, Hyvinkää
  - Päijät-Häme Central Hospital, Lahti

REFERENCES:
- [Derived] Lumikari T, Putaala J, Pirinen J, Kerola A, Sibolt G, Granroth-Wilding H, Pakarinen S, Lehto M, Nieminen T. Empowerment and mobile technology in the detection and treatment of main cardiovascular risk factors of patients with ischemic stroke or transient ischemic attack: a protocol for a multicenter randomized controlled trial (CARDIOSTROKE). Trials. 2025 Mar 14;26(1):89. doi: 10.1186/s13063-025-08778-x. PMID 40082922